CLINICAL TRIAL: NCT07056985
Title: The Effect of Ankle Mobilization Techniques on Balance and Performance in Basketball Players: A Randomized Controlled Clinical Trial
Brief Title: Ankle Mobilization in Basketball Players: Impact on Balance and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Büşra Tamgüç, physiotherapist, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: SBETKK2025-01
Record Dates: First submitted 2025-04-01; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Basketball Players; Mobilization; Jumping Performance
Keywords: basketball players; Mobilization; Jumping Performance

STUDY DESIGN:
Intervention Model Description: This study has a randomized, single-blind, prospective design.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobilization Group (Experimental): Mobilization Group
  Interventions: Other: Ankle joint mobilization technique
- Plasebo group (Placebo Comparator): Plasebo group
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Ankle joint mobilization technique — Combined posterior and lateral mobilization techniques
  Arms: Mobilization Group
Other: Placebo — Placebo interventions simulated with superficial hand contact and minimal manipulation
  Arms: Plasebo group

SUMMARY:
This study aims to evaluate the effects of ankle mobilization techniques on performance in basketball players.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of ankle mobilization techniques on performance in basketball players. The study aims to comparatively reveal the possible effects of mobilization techniques on balance and performance in basketball players.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 24
* Have a body mass index (BMI) ranging from 18.5 kg/m² to 25 kg/m²
* Not have experienced any trunk or lower extremity injuries within the last 6 months prior to the date of participation in the study

Exclusion Criteria:

* Have experienced trunk or lower extremity injuries within the last 6 months prior to the study
* Have a history of fractures or dislocations in the lower extremities
* Have a musculoskeletal system anomaly
* Be unable to perform functional tasks (due to visual, auditory, vestibular, or neurological disorders) (Gahanati et al., 2022)
* Be pregnant
* Have malignancy or metabolic diseases

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Optojump Testing | Participants will be measured with the optojump device twice in total, before and immediately after the intervention.
  The Optojump photocell system is a valid and reliable tool for assessing vertical jump height in both field and laboratory settings. Optojump photoelectric cells (Microgate, Bolzano, Italy) consist of two parallel bars (a receiver and a transmitter unit) placed at ground level. Additionally, the Optojump system offers advantages such as ease of transport and use, as well as being relatively cost-effective (Glatthorn et al., 2011).
Flamingo Balance Test | Participants will be measured with the flamingo balance test twice in total, before and immediately after the intervention.
  The Flamingo Balance Test is one of the most popular field tests for assessing static balance due to its simplicity, low cost, ease of application in various environments, and suitability for large-scale research. In the Flamingo test, the individual stands on one leg on a special wooden beam (50 × 3 × 4 cm) in extension, flexes the free leg at the knee, and holds the foot with the hand on the same side. The evaluator starts the timer as soon as the participant releases the surface they are supporting themselves with. The result is the maximum number of attempts within 1 minute, and this number is limited to 30 (Sember et al., 2020).

CONTACTS AND LOCATIONS:
Locations (1):
- Bahcesehir University, Istanbul, Beşiktaş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided